CLINICAL TRIAL: NCT00311324
Title: A Church Based Intervention to Improve Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 99-0960; U48/CCU409660, 22PR-99 (Other: Centers for Disease Control and Prevention)
Record Dates: First submitted 2006-03-31; First posted 2006-04-05 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2015-12

CONDITIONS: Type 2 Diabetes
Keywords: behavioral intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Special Intervention (Experimental): One individual counseling visit, twelve group sessions, three postcards, and twelve telephone calls.
  Interventions: Behavioral: Special Intervention
- Delayed Intervention (Experimental): Direct mailing of two American Dietary Association pamphlets ("Healthy Eating" and "Staying Alive") and three bimonthly newsletters providing general health information and study updates.
  Interventions: Behavioral: Delayed Intervention

INTERVENTIONS:
Behavioral: Special Intervention
  Other Names: Diabetes self care (behavior)
  Arms: Special Intervention
Behavioral: Delayed Intervention
  Other Names: Diabetes self care (behavior)
  Arms: Delayed Intervention

SUMMARY:
The purpose of this study it to determine if a culturally appropriate, church based intervention for African Americans with type 2 diabetes, will lead to improved glycemic (blood sugar) control.

DETAILED DESCRIPTION:
African Americans suffer disproportionately from diabetes and its complications. To reduce this burden of suffering, innovative interventions are needed to improve self-care behaviors including: dietary intake, physical activity (PA), self-monitoring, and medication adherence. The goal of this study (A New DAWN) was to develop and test a culturally appropriate, church-based intervention to improve diabetes self-management and glycemic control.

Twenty-four African American churches in central NC were recruited and randomized to receive the special intervention (SI-13 churches, 117 participants) or the delayed intervention (DI-11 churches, 84 participants). The SI included an 8-month intensive phase consisting of: 1 individual dietary assessment and counseling visit; 12 group sessions; monthly phone contact with a peer counselor (church diabetes advisor (CDA)); and 3 printed encouragement messages from the primary care clinician. This was followed by a 4-month reinforcement phase including monthly phone contacts from the CDA. At 8- and 12-month follow-up, HbA1c was assessed by high-performance liquid chromatography.

At baseline, 64% of participants were female and means were: age 59, years with diabetes 9, HbA1c 7.8%, Systolic Blood Pressure 139, Diastolic Blood Pressure 76, and BMI 35.0. A total of 174 (87%) participants returned for 8-month measures. Adjusting for baseline values and randomization by church, the mean HbA1c level was 7.4% for the SI and 7.8% for the DI (difference 0.4%, 95% Confidence Interval (CI) 0.1-0.6, p = 0.009). There were no statistically significant differences between groups for BP or BMI. Of 82 (70%) SI participants completing an 8-month follow-up questionnaire, 65 (79%) were very satisfied with the nutritional component, 63 (77%) were very satisfied with the PA component, and 72 (88%) considered the program to be very helpful overall.

In A New DAWN, the SI was acceptable and produced a modest, but clinically significant, reduction in HbA1c. These findings support the acceptability and effectiveness of self-management interventions given in a church setting for African Americans with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* age 20 or older
* diagnosis of type 2 diabetes (diagnosis at age 20 or greater and no history of ketoacidosis)
* clinical care provided by primary care clinician
* plans to reside within 50 miles of church for 1 year
* has home phone or easy access to one

Exclusion Criteria:

* diabetes secondary to another condition
* pregnancy/lactation
* inability to speak English

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2001-02; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Mean Hemoglobin A1c
  5 µL capillary blood collected using standard finger-stick technique and assessed by automated affinity high-performance liquid chromatography.

SECONDARY OUTCOMES:
Mean Dietary recall saturated fat consumption
Median number of minutes per day engaged in physical activity
  Light, Moderate, and Vigorous metabolic equivalents (MET)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Keyserling, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Center for Health Promotion and Disease Prevention/UNC-Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Prev Chronic Disease [serial online] 2006 Jul [date cited]. — http://www.cdc.gov/pcd/issues/2006/jul/05_0085.htm